CLINICAL TRIAL: NCT00463515
Title: A Multicenter Phase II Study of Carboplatin Plus Gemcitabine Followed by Concomitant Chemoradiation in Patients With Non-resectable Stage III Non-Small-Cell-Lung Cancer
Brief Title: Evaluation of Carboplatin Plus Gemcitabine Followed by Concomitant Chemoradiation for Non-resectable Stage III NSCLC
Acronym: CHER@NOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHER@NOS
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Non-Small-Cell-Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Chemoradiation; lung cancer; induction chemotherapy; chemo-radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Gemcitabine; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: carboplatin/gemcitabine
Procedure: cisplatin/radiation therapy

SUMMARY:
The aim of this study is to evaluate whether by combining a carboplatin-gemcitabine based induction chemotherapy with weekly cisplatin during standard thoracic radiotherapy it is possible to obtain optimal efficacy with minimal toxicity. Patients will be treated with 3 cycles of induction chemotherapy, unless there is the occurrence of early intrathoracic progression of disease. The induction chemotherapy is then to be followed by chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* cytological or histologically proven NSCLC
* unresectable stage III NSCLC
* presence of at least one measurable lesion (RECIST criteria)
* adequate haematological, renal and hepatic function
* adequate lung function reserve
* good condition, weight loss <10% over previous 6 months, life expectancy > 3 months

Exclusion Criteria:

* previous chemotherapy for NSCLC
* distant metastasis or a pleural or pericardial effusion
* treatment for malignant disease in the past or serious concomitant medical or psychiatric disease
* active uncontrolled infection at time of inclusion
* interstitial lung disease
* auto-immune systemic disease with potential involvement of the lungs
* concomitant use of amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77
Dates: Start 2003-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
2-year survival rates

SECONDARY OUTCOMES:
Response rate
Time to intrathoracic failure
Overall survival
Toxicity of induction chemotherapy
Toxicity of chemo-radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Germonpre, Principal Investigator — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - ZNA Middelheim, Antwerp, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - Sint Augustinus Ziekenhuis, Wilrijk, Antwerp